CLINICAL TRIAL: NCT07324577
Title: Effectiveness of Virtual Reality in the Management of Anxiety for Patients Undergoing Radiotherapy
Brief Title: Effectiveness of Virtual Reality (VR) in the Management of Anxiety for Patients Undergoing Radiotherapy
Acronym: RELAX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Wake Forest Baptist (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00140668; ONC-LUN-2407 (Other: Atrium Health Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2025-11-18; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Radiation Therapy; Virtual Reality
Keywords: Virtual Reality; Cancer; Radiation Therapy
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (Other): Standard of care radiation therapy for prostate, lung, breast cancer without using the VR headset
  Interventions: Other: standard of care
- Virtual Reality intervention (Other): Participants will wear the VR headset (Quest 2 by Meta) during radiation therapy
  Interventions: Other: standard of care; Other: Virtual Reality Intervention
- Radiation Therapists (Other): Providers that administer the VR intervention
  Interventions: Other: Radiation Therapist Survey

INTERVENTIONS:
Other: standard of care — Radiation therapy for prostate cancer, breast cancer, lung cancer, or head and neck cancer.
  Arms: Standard of care; Virtual Reality intervention
Other: Virtual Reality Intervention — Participants will wear the VR headset (Meta Quest 2) during standard of care radiation therapy
  Arms: Virtual Reality intervention
Other: Radiation Therapist Survey — Radiation therapists will be asked about their experiences and proficiency with using the VR device.
  Arms: Radiation Therapists

SUMMARY:
The purpose of this study is to evaluate the use and functionality of virtual reality (VR) during radiation therapy treatments for patients with prostate, breast, lung, or head and neck cancer.

DETAILED DESCRIPTION:
This is a randomized controlled trial that will assess the feasibility, acceptability, tolerability, and initial clinical efficacy of using a VR device during radiation therapy for participants with prostate cancer, breast cancer, lung cancer, or head and neck cancer.

Participants will be randomized 2:1 to either the VR device intervention arm or the standard of care control arm.

Participants will undergo pre-study assessments, assessments before and after the first radiation treatment, every 6th radiation treatment, and at the end of treatment.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Participants planned for radiation therapy for 15 or more treatments with non-neutron generating energies (10 MV or less) per study PI for prostate, breast, lung, or head and neck cancer. Neutrons have the potential to damage the VR headset device and are generated for energies above 10 MV.
* Age 18 years or older at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3 at the time of enrollment.
* Ability to understand and the willingness to sign an IRB-approved informed consent document directly.

Exclusion Criteria:

* Previous radiation therapy
* VR device is determined to impede the radiation dosage during the VR device simulation and treatment planning
* Participants with primary brain tumors, brain metastases, and cancer involving the sinuses, orbits, nose, or ears, are excluded from this clinical trial because the VR device may obstruct the area being treated
* Participants with uncontrolled inter-current illness including but not limited to psychiatric illness/social situations that would limit compliance with study requirements per treating radiation oncologist.
* Participants with known epilepsy, significant motion sickness, severe uncorrected visual impairment, severe uncorrected hearing impairment, or seizures, per participant report.
* Participants with skin defects, infections, or open wounds in the area where the VR device is applied (face or scalp) or in the eyes per treating radiation oncologist.
* Participants with pacemakers, internal defibrillators, hearing aid, or other implanted medical device. The Meta Quest device contains magnets and components that emit magnetic/electromagnetic fields which could affect the operation of nearby electronics and medical devices.

Radiation Therapists:

Inclusion Criteria:

* Agreement to participate after reviewing the information sheet
* Radiation therapist at AHWFBCCC High Point who has treated at least one participant who enrolled on to the study and used the VR device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
VR Use During Treatment | Periprocedural (each treatment visit)
  A binary variable (Yes/No) will be created for participants at the level of individual treatment visit to signify whether the participants wore the VR device for the duration of their treatment.
VR Functionality | Periprocedural (each treatment visit)
  VR device functionality (0-2) will be determined at the level of individual treatment visit using the following criteria as determined by the participant and/or treatment staff:
  0 = device not functional at any time during the treatment
  1. = device functional for part but not all of the treatment duration
  2. = device was functional for the duration of the treatment

SECONDARY OUTCOMES:
Anxiety - Change over time | GAD-7: Baseline RTEQ: Periprocedural (After first and last treatment)
  Generalized Anxiety Disorder 7-item (GAD-7) to assess pre-existing generalized anxiety and the 23-item Radiotherapy Experience Questionnaire (RTEQ) situational unease and situational repose subscales.
Acceptability of Implementing VR | At 36 months
  Radiation Therapist Survey (Administered to staff only)

OTHER OUTCOMES:
Incidence of Treatment - Treatment Related Adverse Events | Periprocedural (each treatment visit)
  Total counts and grade of symptoms such as nausea, dizziness, seizures, blurred vision, fatigue, eye or muscle twitching, instability in posture, blackouts triggered by light flashes or patterns, and headache.
Anxiety - Change over the course of treatment | Periprocedural (first treatment, last treatment, weekly during treatment)
  Single Item Anxiety Questionnaire
Anxiety - Change over the course of treatment | Periprocedural (first treatment, last treatment, weekly during treatment)
  Anxiety evaluation with heart rate
Participant Satisfaction | 4-6 weeks following randomization
  VR Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Parker, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist Hayworth Cancer Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No